CLINICAL TRIAL: NCT02078167
Title: Long Term Efficacy and Tolerability of a Nutraceutical Combination (Red Yeast Rice, Policosanols and Berberine) in Low-moderate Risk Hypercholesterolemic Patients: a Double-blind, Placebo Controlled Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Comitato Etico di Area Vasta Sud Est (Other)
Collaborators: Carla Caffarelli (Unknown)
Responsible Party: Principal Investigator, Stefano Gonnelli, Stefano Gonnelli, Comitato Etico di Area Vasta Sud Est
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ARMOLIPID
Record Dates: First submitted 2014-03-03; First posted 2014-03-05 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Hypercholesterolemia
Keywords: ipercholesterolemia not familiarity
MeSH Terms: conditions — Hypercholesterolemia | interventions — red yeast rice; Berberine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: nutraceutical combination (red yeast rice, policosanols and berberine)
  Other Names: ARMOLIPID

SUMMARY:
Background: Statins are at the forefront of strategies to manage hypercholesterolemia. However, 10-15% of patients result to be intolerant to any statins, even at low daily doses and almost one- third of statin users discontinue therapy within one year. Some nutraceuticals are prescribed as lipid- lowering substances, but doubts remain about their efficacy and tolerability. In this study we investigated the effects of a nutraceutical combination consisting mainly of red yeast rice extract 200 mg (equivalent to 3 mg monacolins), berberine 500 mg and policosanols 10 mg (MBP-NC).

Methods: In this single centre, randomized, double-blind, placebo-controlled study 60 consecutive outpatients (age range: 18-60 years), with newly diagnosed primary hypercholesterolemia not previously treated, after a run-in period of 3 weeks on a stable hypolipidic diet, were randomized to receive a pill of MBP-NC (N=30) or placebo (N=30) once a day after dinner, in addition to the hypolipidic diet. The efficacy and the tolerability of the proposed nutraceutical treatment were fully assessed after 4, 12 and 24 weeks of treatment.

DETAILED DESCRIPTION:
Introduction Many epidemiological studies have shown that serum cholesterol levels are strongly related to cardiovascular risk [1, 2]. Consequently lowering cholesterol levels is a fundamental prognostic goal in the primary and secondary prevention of cardiovascular events. The 3-hydroxy-3-methylglutaryl-coenzime A (HMG-CoA) reductase inhibitors, commonly known as "statins" are at the forefront of strategies to manage hypercholesterolemia, especially in patients at high or very high risk of cardiovascular diseases, in view of their established efficacy in reducing cardiovascular mortality and morbidity in both primary and secondary prevention [3, 4]. However, 10-15% of patients result to be intolerant to any statins, even at low daily doses and almost one-third of statin users discontinue therapy within one year from the beginning [4, 5]. Furthermore, the use of statins to reduce cardiovascular risk in clinical practice is rarely encouraged for primary prevention and some other patients, especially in primary prevention, refuse statins because of the fear of possible side effects. Some nutraceutical products may represent an alternative treatment to be considered for the above mentioned cases, above all in patients with marginally high hypercholesterolemia [4, 6]. Since the use of full- dose nutraceuticals entails some tolerability concerns, a combination of nutraceuticals with different but synergic mechanisms of action at lower and safer dosages could be preferable. In particular, in recent years there has been a growing interest in a nutraceutical combination containing monakolin (the biologically active component of red yeast rice), berberine and policosanols (MBP-NC). The cholesterol lowering effect of MBP-NC consumed in conjunction with a standard Mediterranean healthy diet has been observed in a large Italian study carried out by general practitioners (GPs) [7], in patients intolerant to more than one statin [8], in patients with metabolic syndrome or who are overweight [9, 10] and in elderly hypercholesterolemic subjects [11]. Moreover, MBP-NC mixture has been reported to have some direct protective vascular effects, similar to pharmacological lipid lowering agents, such as improvement in endothelial dysfunction [12] and improvement in aortic stiffness [13]. Another recent study has reported that a 2-month treatment with MBP-NC improved insulin sensitivity in patients with metabolic syndrome [14].

However, hitherto the cholesterol lowering effect of MBP-NC has not been evaluated in long term double-blind placebo controlled studies. The aim of this single centre, randomized, double-blind, placebo-controlled study was to evaluate the efficacy and the safety of a 24 week treatment with MBP-NC mixture in low -moderate risk hypercholesterolemic patients.

Materials and Methods Population A cohort of 66 consecutive outpatients with newly diagnosed primary hypercholesterolemia not previously treated who applied to the Lipid Clinic of the Department of Internal Medicine at the University of Siena (Italy), were considered for enrolment in this study. The inclusion criteria were (1) age between 18 and 60 years , (2) body mass index(BMI) between 18,5 ad 29,9 Kg/m2, (3) serum low-density lipoprotein cholesterol (LDL-C) above 150 mg/dL and an estimated 10-year cardiovascular risk < 20% according to Framingham risk scoring. The exclusion criteria were (1) history of cardiovascular disease or coronary risk equivalents, (2) secondary hyperlipidemia caused by diabetes mellitus, renal, liver or thyroid diseases, (3)alcohol consumption of > 40 g/day, (4) estimated 10-year cardiovascular risk > 20% according to Framingham risk scoring, (5) muscular diseases or abnormally elevated creatine phosphokinase (CPK) levels or drug treatment with anti-platelet, anti-inflammatory, hypolipidemic agents or hormone replacement therapy, either on-going or any time in the previous 2 months. Instead, the patients on stable anti-hypertensive treatment for at least 3 months were included. All the patients were instructed to maintain their habitual physical activity during the study period.

At the screening visit, all patients were instructed to follow a hypolipidic diet (low- cholesterol/ low-saturated fat diet approximately consisting of 55% carbohydrates, 20% proteins, and 25% lipids) during a run-in period of 3 weeks, after which all patients who met the inclusion criteria, were randomized to receive a pill of MBP-NC (N=30 ) or placebo (N=30) once a day after dinner, in addition to the hypolipidic diet. The placebo pills, identical in taste and appearance to the MBP-NC pills, consisted of inactive compound. Randomisation and blinding were provided by Rottapharm Madaus S.p.A (Monza, Italy). The composition of the patented proprietary combination of nutraceuticals investigated was as follows: red yeast rice extract 200 mg (equivalent to 3 mg monacolins), berberine 500 mg, policosanol 10 mg, folic acid 0.2 mg, coenzyme Q10 2 mg and asthaxantin 0.5 mg (Armolipid Plus, Rottapharm Madaus S.p.A, Italy).

The study was conducted in accordance with the guidelines of the Declaration of Helsinki, as revised in 2000 and 2008, and the study protocol was approved by the Ethics Committee of the University Hospital of Siena. Written informed consent was obtained from each patient.

Clinical and anthropometric evaluation All patients underwent physical examination at baseline and after 4, 12, and 24 weeks of treatment. All the determinations were made at the Lipid Clinic at 09.00 AM , after an overnight fast of 12 h. Height and weight were measured to the nearest 0.1 cm and 0.1 Kg, respectively. BMI was calculated as weight in kilograms divided by height squared in meters. Brachial blood pressure was measured by a physician with a mercury sphygmomanometer after patient had been seated for at least 10 min and the average of 3 measurements was considered for the analysis. Waist circumference was also measured at each visit midway between the lowest rib and the iliac crest using an anthropometric tape.

In all patients, body composition [fat mass (FM) percentage, fat-free mass (FFM) and fat-free mass/fat mass ratio (FFM/FM)] was assessed by anthropometry and bioelectrical impedance analysis (BIA) using a single-frequency 50 kHz bioelectrical impedance analyzer (BIA 101 RJL, Akern Bioresearch, Florence, Italy). All BIA measurements were carried out by the same operator according to the standard tetrapolar technique, with patients in a supine position for at least 20 min. The electrodes were placed on the dorsal surface of the right foot and ankle and the right wrist and hand. Biochemical measurements In all patients fasting venous blood samples were drawn at baseline and after 4, 12 and 24 weeks in order to assess serum levels of total cholesterol (TC), triglycerides (TG), high-density lipoprotein cholesterol (HDL-C) and low-density lipoprotein cholesterol (LDL-C). All lipid parameters (TC, TG, HDL-C and LDL-C) were measured using a colorimetric method (Autoanalyzer Menarini, Florence, Italy). In order to monitor the safety of the MBP-NC in all patients, at the same time points, serum levels of glucose, uric acid, CPKw, gammaglutamiltranferase (ɣGT) and transaminases were also assessed. Tolerability was monitored by recording symptoms. Medication compliance was assessed by counting the number of pills returned at the clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were (1) age between 18 and 60 years , (2) body mass index(BMI) between 18,5 ad 29,9 Kg/m2, (3) serum low-density lipoprotein cholesterol (LDL-C) above 150 mg/dL and an estimated 10-year cardiovascular risk < 20% according to Framingham risk scoring.

Exclusion Criteria:

* The exclusion criteria were (1) history of cardiovascular disease or coronary risk equivalents, (2) secondary hyperlipidemia caused by diabetes mellitus, renal, liver or thyroid diseases, (3)alcohol consumption of > 40 g/day, (4) estimated 10-year cardiovascular risk > 20% according to Framingham risk scoring, (5) muscular diseases or abnormally elevated creatine phosphokinase (CPK) levels or drug treatment with anti-platelet, anti-inflammatory, hypolipidemic agents or hormone replacement therapy, either on-going or any time in the previous 2 months.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
level of cholesterol | 24 weeks
level of tryglicerides | 24 weeks

REFERENCES:
- [Derived] Gonnelli S, Caffarelli C, Stolakis K, Cuda C, Giordano N, Nuti R. Efficacy and Tolerability of a Nutraceutical Combination (Red Yeast Rice, Policosanols, and Berberine) in Patients with Low-Moderate Risk Hypercholesterolemia: A Double-Blind, Placebo-Controlled Study. Curr Ther Res Clin Exp. 2014 Nov 15;77:1-6. doi: 10.1016/j.curtheres.2014.07.003. eCollection 2015 Dec. PMID 26649075